CLINICAL TRIAL: NCT00637052
Title: A Phase 1/2 Study of ARRY-520 in Patients With Advanced Myeloid Leukemia
Brief Title: A Study of ARRY-520 in Patients With Advanced Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: ARRAY-520-211; C4371005 (Other: Alias Study Number)
Record Dates: First submitted 2008-02-22; First posted 2008-03-17 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Advanced MDS; Acute Myeloid Leukemia
Keywords: preleukemia; dysplasia of myeloid blood cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Preleukemia | interventions — filanesib

ARMS (1):
- ARRY-520 (Experimental)
  Interventions: Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous

INTERVENTIONS:
Drug: ARRY-520, KSP(Eg5) inhibitor; intravenous — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule; Part 3: multiple dose, single schedule.

SUMMARY:
This is a 2-phase study during which patients with select myeloid leukemias or advanced myelodysplastic syndrome (MDS), who have failed, refused or are not eligible for standard treatment, will receive investigational study drug ARRY-520.

The study has 3 parts. The first phase of the study, Phase 1, has 2 parts. In the first part of Phase 1, patients with select myeloid leukemias or advanced MDS will receive increasing doses of study drug on different schedules in order to achieve the highest dose possible that will not cause unacceptable side effects. Approximately 30 patients (per schedule) from the US will be enrolled in Part 1 (Completed). In the second part of Phase 1, patients with advanced MDS will receive the best dose of study drug and schedule determined from the first part of the study. Approximately 10 patients from the US will be enrolled in Part 2 (Completed).

In the third part of the study, Phase 2, patients with acute myeloid leukemia (AML) or advanced MDS will receive the best dose of study drug and schedule determined from the first part of the study and will be followed to see what side effects the study drug causes and to see what effectiveness it has, if any, in treating the cancer. Approximately 40 patients from the US will be enrolled in Part 3 (Withdrawn).

ELIGIBILITY:
Key Inclusion Criteria (Part 2):

* Patients with either Intermediate-2 or High risk MDS or with AML (>20% bone marrow blasts) with stable low or normal white blood cell count (WBC). Patients should have failed one prior chemotherapy regimen which should have included a hypomethylating agent.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Discontinuation of prior treatment at least 2 weeks prior to the start of the study.
* Adequate hepatic and renal function.
* Additional criteria exist.

Key Exclusion Criteria (Part 2):

* Concurrent cytotoxic therapy, or biological, endocrine and immunological response modifiers.
* Previous radiation to >25% of bone marrow.
* Other active malignancies.
* Known positive serology for the human immunodeficiency virus (HIV).
* Central nervous system involvement as documented by spinal fluid cytology.
* Active, uncontrolled infection.
* Additional criteria exist

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03-18 (Actual); Primary Completion 2010-06-21 (Actual); Study Completion 2010-06-21 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of the study drug. | Part 1
Characterize the pharmacokinetics (PK) of the study drug. | Part 1
Characterize the safety profile of the study drug in terms of adverse events, dose limiting toxicity, clinical laboratory tests, weight, electrocardiograms and physical examinations. | Part 1 and Part 2
Assess the efficacy of the study drug in terms of incidence of complete remission (CR) and hematologic improvement (CRp). | Part 3

SECONDARY OUTCOMES:
Assess the efficacy of the study drug in terms of incidence of CR and CRp. | Part 1 and Part 2
Characterize the safety profile of the study drug in terms of adverse events, dose limiting toxicity, clinical laboratory tests, weight, electrocardiograms and physical examinations. | Part 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Emory University School of Medicine, Winship Cancer Center, Atlanta, Georgia
  - University of Texas, M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Khoury HJ, Garcia-Manero G, Borthakur G, Kadia T, Foudray MC, Arellano M, Langston A, Bethelmie-Bryan B, Rush S, Litwiler K, Karan S, Simmons H, Marcus AI, Ptaszynski M, Kantarjian H. A phase 1 dose-escalation study of ARRY-520, a kinesin spindle protein inhibitor, in patients with advanced myeloid leukemias. Cancer. 2012 Jul 15;118(14):3556-64. doi: 10.1002/cncr.26664. Epub 2011 Dec 2. PMID 22139909